CLINICAL TRIAL: NCT00946478
Title: A Three-week, Double-blind, Randomized Study to Evaluate the Effect of Pimecrolimus Cream 1% on Cathelicidin Expression in the Skin of Subjects With Atopic Dermatitis
Brief Title: Effect of Pimecrolimus Cream on Cathelicidin Levels in Subjects With Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Richard Gallo, Chair, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCSDMED
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-01

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; elidel; pimecrolimus; CASM981; immunity; cathelicidin; antimicrobial peptide; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pimecrolimus (Active Comparator)
  Interventions: Drug: Pimecrolimus
- Vehicle cream (Sham Comparator)
  Interventions: Other: Vehicle cream

INTERVENTIONS:
Drug: Pimecrolimus — 20 AD patients will be given pimecrolimus 1% to apply twice daily for up to three weeks on each lesional site predetermined at baseline. Lesional target site and non-lesional site will be determined at Visit 1.
  Two 2 mm biopsies will be obtained from a target AD lesion and non-lesional sites at Visit 2, and Visit 3 (four biopsies each visit).
  Other Names: Elidel; CASM 981
  Arms: Pimecrolimus
Other: Vehicle cream — 20 AD patients will be treated with vehicle cream twice daily for up to 3 weeks on each lesional site predetermined at baseline. Lesional target site and non-lesional site will be determined at Visit 1.
  Two 2 mm biopsies will be obtained from a target AD lesion and non-lesional sites at Visit 2, and Visit 3 (four biopsies each visit).
  Arms: Vehicle cream

SUMMARY:
The purpose of this study is to determine the effect of topical pimecrolimus on the immune system by assessing the levels of antimicrobial peptides in the skin of patients with eczema. It is hypothesized that pimecrolimus applied topically will repair the body's immune system in patients with eczema by increasing antimicrobial peptides.

DETAILED DESCRIPTION:
Patients with atopic dermatitis (AD) have higher rates of skin infections from viruses and bacteria. They also have an impaired innate immune system. Antimicrobial peptides are a component of the innate immune system which are decreased in atopics. In vitro, pimecrolimus has demonstrated its ability to increase antimicrobial peptides. This study will examine the ability of pimecrolimus to increase antimicrobial peptides in vivo in AD patients. Thus, the study will yield a better understanding of the role of pimecrolimus in regulating the immune system in atopics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Target lesion IGA ≥2
3. Target IGA=0 (for non-lesional site)
4. Male or female of any race and ethnicity
5. Chronic AD for more than one year duration
6. Subject of child-bearing potential must be willing to practice effective birth control during the study
7. Subject agrees to comply with study requirements and attend all required visits.

Exclusion Criteria:

1. Patients ≥ 18 years of age with only AD of the face
2. Women of childbearing potential not using the contraception method(s) specified in this study (abstinence, IUD, diaphragm, oral contraceptives)
3. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
4. Hypersensitivity to pimecrolimus cream or any excipient of the cream
5. Subject has a skin disorder in addition to dermatitis in the areas to be treated
6. Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
7. Pregnant or nursing females
8. Immunocompromised patient (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or with a history of active or malignant disease (excluding non-melanoma skin cancer)
9. History of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
10. Patients known to be non-compliant with a medication regimen
11. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
12. Active viral or fungal skin infections at the target areas
13. Previous participation in this study
14. Ongoing participation in another investigational trial
15. Use of any oral or topical antibiotic during the study and up to one week prior to entering the study
16. Use of any local therapy for AD less than one week prior to screening
17. Use of any systemic immunosuppressive therapy for AD less than four weeks prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego - Dept of Dermatology, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimecrolimus: Pimecrolimus: 20 AD patients will be given pimecrolimus 1% to apply twice daily for up to three weeks on each lesional site predetermined at baseline. AD severity will be evaluated by the Investigator Global Assessment of Disease Activity (IGA). The IGA scale is 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe disease. The patient's AD will be evaluated on Visit 1 (Day -14 to 1), Visit 2 (Day 1), and Visit 3 (Week 21). Lesional target site and non-lesional site will be determined at Visit 1.
  Two 2 mm biopsies will be obtained from a target AD lesion and non-lesional sites at Visit 2, and Visit 3 (four biopsies each visit).
- Vehicle Cream: Vehicle cream: 20 AD patients will be treated with vehicle cream twice daily for up to 3 weeks on each lesional site predetermined at baseline. AD severity will be evaluated by the Investigator Global Assessment of Disease Activity (IGA). The IGA scale is 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe disease9. The patient's AD will be evaluated on Visit 1 (Day -14 to 1), Visit 2 (Day 1), and Visit 3 (Week 21). Lesional target site and non-lesional site will be determined at Visit 1.
  Two 2 mm biopsies will be obtained from a target AD lesion and non-lesional sites at Visit 2, and Visit 3 (four biopsies each visit).
Period: Overall Study
Arm/Group | Pimecrolimus | Vehicle Cream
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimecrolimus | Vehicle Cream | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (8.4) | 28.6 (9.5) | 27.4 (9)
Sex/Gender, Customized [Number; unit: participants] — Gender
  participants
    Male | 9 | 6 | 15
    Female | 7 | 7 | 14
    Unknown | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cathelicidin mRNA Expression Levels in Adult Skin From Patients With AD
Description: Delta-delta CT values were measured using RT-PCR of cathelicidin mRNA in human biopsy samples at baseline, and then 3 weeks after treatment with either pimecrolimus or placebo
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: delta-delta ct units on PCR
Arm/Group | Pimecrolimus | Vehicle Cream
Number analyzed (Participants) | 20 | 20
delta-delta ct units on PCR | .0016 (.002) | .0024 (.004)

ADVERSE EVENTS:
Arm/Group | Pimecrolimus | Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes